CLINICAL TRIAL: NCT05041933
Title: Pilot Study: Secure Outsourcing of Carfilzomib in the Treatment of Multiple Myeloma to the Hospital at Home (HAH) Setting. Care Organisation Model for New Short Intravenous Infusion Chemotherapies
Brief Title: Secure Outsourcing of Carfilzomib in the Treatment of Multiple Myeloma to the Hospital at Home Setting
Acronym: Carfil-HAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20_0054
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-08

CONDITIONS: Hematological Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: outsourcing of chemotherapy to Hospital at Home — outsourcing of chemotherapy to Hospital at Home

SUMMARY:
Since 2009, the Department of Clinical Haematology at Limoges University Hospital Centre, supported by the HEMATOLIM network, has been operating the regional "ESCADHEM" system: [Secure outsourcing of injectable chemotherapy to the home care setting for malignant blood diseases]. In addition to Limoges University Hospital, Brive Hospital and Guéret Hospital, this system involves four Hospital at Home (HAH) structures across the three départements of the former Limousin region.

In this process, chemotherapy administered by subcutaneous injection is prescribed by a hospital physician in one of the hospitals "authorised to deliver cancer treatments" in the former region of Limousin: Limoges University Hospital Centre, Brive Hospital or Guéret Hospital. This chemotherapy is then prepared in one of the three hospital pharmacies authorised to perform centralised reconstitution, in accordance with current standards. The preparation is then transferred to one of the four Hospital at Home (HAH) structures, which transports the product to the patient's home where it is administered by the nurse (IDE). This last step in the process is under the responsibility of the HAH structure coordinating physician, who is also responsible for waste collection.

Supported by its experience within the ESCADHEM system with subcutaneous drugs and in the context of the arrival of new intravenous drugs, in short infusion form, the Department of Clinical Haematology, supported by the HEMATOLIM network (which became the HEMATOLIM association on 1 January 2020) and the professionals involved began the process of outsourcing these drugs to the HAH setting. One of these drugs is carfilzomib, used to treat multiple myeloma, and its outsourcing to the HAH setting was put in place from the end of 2018.

In parallel with this, the Department of Clinical Haematology would like to set up a study to evaluate the feasibility of outsourcing this new drug, administered intravenously, based on a model that we know to be operational and secure for chemotherapies administered by subcutaneous injection.

the Department of Clinical Haematology hope to be able to confirm the value of caring for multiple myeloma patients in an HAH setting by improving their quality of life and optimising their care pathway in organisational and economic terms. the Department of Clinical Haematology hope to be able to demonstrate that this organisation is not only efficient in the view of patients, but also for the healthcare professionals working in the Hospital, the HAH structure and in the community, involved throughout the care process.

To conduct our study, the Department of Clinical Haematology selected the novel drug carfilzomib, used in the treatment of multiple myeloma.

The prescribing conditions, treatment administration regimen and outsourcing quality processes for this drug are available in the annexes. These standard regimens were constructed on the basis of the protocols in the ESCADHEM system, extensively trialled and validated by the HAS, for drugs injected subcutaneously and following a collegial approach. We thus hope to demonstrate that the protocols used for drugs administered by subcutaneous injection - in particular, bortezomib and azacytidine - are applicable to carfilzomib following minor modifications to the procedures given the IV administration of the latter drug as a short infusion.

It should be noted that it is essential that the first cycle of carfilzomib be administered, in its entirety, in an outpatient clinic setting. Thereafter, if the patient is eligible for treatment in an HAH setting, the 1st day of each cycle will be performed in an outpatient clinic.

Following this study, the Department of Clinical Haematology hope to be able to publish our research and promote it at national and/or international congresses. This research should further reinforce our already significant experience in this type of care strategy for malignant blood diseases in the HAH setting, which we believe is simultaneously innovative, practical and beneficial for all the players in the care pathway concerned. The model will probably be useful for outsourcing to the HAH setting other novel drugs progressively arriving on the market with profiles similar to that of the drug we wish to study.

Finally, our project aims to demonstrate that our procedures for the secure outsourcing of carfilzomib to the HAH setting, in place since the end of 2018 are valid and could be extended to other regions of France. Furthermore, the current health landscape is undergoing profound changes associated with budget constraints, as well as societal and technological evolutions, with the result that home care, and hence HAH structures, appear, more than ever, to be the model of the future.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or over.
* Eligible for care by one of the four HAH structures in accordance with HAS criteria,
* With relapsed or refractory multiple myeloma (having received at least one previous treatment),
* Whose case has been examined at multidisciplinary team (MDT) meetings at Limoges University Hospital Centre,
* Receiving carfilzomib parenteral chemotherapy outsourced to an HAH setting (all patients receive the entire first cycle of carfilzomib and the 1st day of each of the subsequent cycles in an outpatient clinic).
* Having read the information leaflet concerning the Carfil-HAD study,
* Not objecting to the use of their data in the context of this study.

Exclusion Criteria:

* Inability to understand the protocol or complete the questionnaires.
* Refusing to complete the questionnaires.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with relapsed or refractory multiple myeloma (having received at least one previous treatment),
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Number of deviations from SOPs occurring in the context of secure outsourcing of carfilzomib administered by short IV infusion, for 3 cycles, to a mixed outpatient clinic/HAH care setting. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No